CLINICAL TRIAL: NCT03589833
Title: Effectiveness and Safety of Tumor Necrosis Factor Receptor Fusion Protein(Yisaipu) Combined With Tripterygium Wilfordii for Active Rheumatoid Arthritis
Brief Title: Effectiveness and Safety of Yisaipu Combined With Tripterygium Wilfordii for Active RA
Acronym: YISTAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xuan Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YISTAR
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Methotrexate; Tripterygium; TNF inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MTX (Placebo Comparator): Treated with oral methotrexate and two placebos.
  Interventions: Drug: Methotrexate
- Tripterygium Wilfordii (Placebo Comparator): Treated with oral Tripterygium Wilfordii and two placebos.
  Interventions: Drug: Tripterygium Wilfordii
- Yisaipu + MTX (Active Comparator): Treated with subcutaneously injected Yisaipu, oral methotrexate and a placebo.
  Interventions: Drug: Methotrexate; Drug: Yisaipu
- Yisaipu + Tripterygium Wilfordii (Experimental): Treated with subcutaneously injected Yisaipu, oral methotrexate and a placebo.
  Interventions: Drug: Tripterygium Wilfordii; Drug: Yisaipu

INTERVENTIONS:
Drug: Tripterygium Wilfordii — Oral Tripterygium Wilfordii 20mg thrice daily for 24 weeks.
  Arms: Tripterygium Wilfordii; Yisaipu + Tripterygium Wilfordii
Drug: Methotrexate — Oral methotrexate 7.5-15mg per week for 24 weeks. The starting dose was 7.5mg per week, then increased to 15mg (max 0.3mg/Kg) per week in 4 weeks. Folic acid at the dose of 5 mg per week were applied to all participants.
  Arms: MTX; Yisaipu + MTX
Drug: Yisaipu — Yisaipu, a Tumor Necrosis Factor Receptor Fusion Protein, was subcutaneously injected at a dose of 50 mg once a week for 24 weeks.
  Arms: Yisaipu + MTX; Yisaipu + Tripterygium Wilfordii

SUMMARY:
In this 24-week, multi-center, randomized, double-blind study, the investigators will evaluate the efficacy and safety profile of subcutaneously injected Yisaipu, a Tumor Necrosis Factor Receptor Fusion Protein, combined with oral Tripterygium Wilfordii for patients with active rheumatoid arthritis.

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of YISAIPU plus Tripterygium wilfordii (T2w) for the treatment of RA patients. YISAIPU is a recombinant human tumor necrosis factor receptor fusion protein, and tripterygium wilfordii is a chloroform/methanol extract of Tripterygium wilfordii Hook F.

Objectives:

1. To compare the efficacy of YISAIPU plus T2w versus MTX monotherapy for the treatment of signs and symptoms of RA.
2. To evaluate the safety of YISAIPU plus T2w in patients with RA for 24 weeks.

Design:

This is a randomized, 24-week, double-blind, parallel group study, and 506 patients with active RA will be randomized in a 1:1:1:1 ratio to one of the following four parallel treatment arms:

1. Methotrexate monotherapy
2. T2w monotherapy
3. YISAIPU plus methotrexate
4. YISAIPU plus T2w

Escape:

On week 13, all participants with inadequate response, defined as a <30% improvement of swollen and tender joint counts from baseline, will switch to YISAIPU plus T2w treatment throughout the study.

Endpoints :

1. ACR20, ACR50 and ACR70 response rates at 12 and 24 weeks.
2. DAS 28 (CRP) and DAS 28 (ESR) at 12 and 24 weeks.
3. EULAR response rates at 12 and 24 weeks.
4. Health assessment questionnaire (HAQ) at 12 and 24 weeks.
5. Patient assessment of arthritis pain at 12 and 24 weeks.
6. Patient and physician global assessment of arthritis at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years with informed consent
* Diagnosis of rheumatoid arthritis (according to 2010 ACR/EULAR classification criteria)
* Disease duration > 6 weeks
* Swollen joint (SJC)≥4 and tender joint count(TJC)≥4
* ESR >28 mm/hr or C-reactive protein > 1.5 ULN
* Positive RF or anti-CCP antibody on screening
* Class I, II or III of the ACR 1991 Revised Criteria for Global Functional Status in RA
* No evidence of active or latent or inadequately treated Mycobacterium tuberculosis infection

Exclusion Criteria:

* Pregnant, lactating or further fertility requirements
* Previously received any biologic agents.
* Recently (<12 weeks) received methotrexate, leflunomide, salazosulfapyridine, azathioprine, cyclosporine, mycophenolate mofetil or Tripterygium Wilfordii.
* Active or chronic infection, including HIV, HCV, HBV, tuberculosis.
* History of any other rheumatic autoimmune disease
* History of any lymphoproliferative disorder
* Malignancy or history of malignancy.
* Abnormal laboratory tests, including: Hemoglobin <8.5 g/dL, White blood cell count <3.5 x 109/L, Platelet count <100 x 109/L, AST/ALT >1.5 ULN, and serum creatine > 1.5 mg/dL.
* Severe, progressive, or uncontrolled cardiac, pulmonary, renal, hepatic, gastrointestinal, hematologic, metabolic, endocrine or neurologic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
The American College of Rheumatology 50 (ACR50) response at 12 weeks | week 12
  The difference of ACR50 between Arm 4 (Yisaipu + Tripterygium Wilfordii) and Arm 1 (MTX) at week 12.

SECONDARY OUTCOMES:
The American College of Rheumatology 20/70 (ACR20/ACR70) response at 12 weeks | week 12
  The difference of ACR20 and ACR70 between Arm 4 (Yisaipu + Tripterygium Wilfordii) and Arm 1 (MTX) at week 12.
The American College of Rheumatology 20/50/70 (ACR20/ACR50/ACR70) response at 24 weeks | week 24
  The difference of ACR20, ACR50 and ACR70 between Arm 4 (Yisaipu + Tripterygium Wilfordii) and Arm 1 (MTX) at week 24.
The Disease Activity Score-28 (DAS28) response at 24 weeks | week 24
  The change in DAS28 score from baseline to week 24 between Arm 4 (Yisaipu + Tripterygium Wilfordii) and Arm 1 (MTX).
  DAS28 ＝ 0.56*SQRT(TJC28) + 0.28*SQRT(SJC28) + 0.36*ln(CRP + 1) + 0.014*GH + 0.96
  * TJC28: The number of tender joints (0-28).
  * SJC28: The number of swollen joints (0-28).
  * CRP: The C-Reactive Protein level (in mg/l).
  * GH: The patient global health assessment (from 0=best to 100=worst).
  The 28 joint: shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees.
The European League Against Rheumatism (EULAR) response at 12 weeks | week 12
  The difference of proportions of patients meeting EULAR response between Arm 4 (Yisaipu + Tripterygium Wilfordii) and Arm 1 (MTX) at week 12.
Health Assessment Questionnaire without Didability Index (HAQ-DI) at 12 weeks | week 12
  The change in HAQ-DI score from baseline to week 12 between Arm 4 (Yisaipu + Tripterygium Wilfordii) and Arm 1 (MTX).
  HAQ-DI is an index measuring the quality of life related to health, which includes 20 questions in terms of three categories:
  * from 0 to 1: mild difficulties to moderate disability,
  * from 1 to 2: disability moderate to severe,
  * from 2 to 3: severe to very severe disability.
  The mean score is recorded as the result.

OTHER OUTCOMES:
The Incidence of adverse events during 24-week study | week 24
  Incidence of adverse events and sever adverse events (SAE), including hospitalized or Treatment-emergent adverse events, during 24-week study.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Deptment of Rheumatology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang X, Yang H, Zuo X, Wu L, Peng J, Li Z, Li H, Ji W, Zhang L, Li X, Dai L, Lu L, Yang N, Wei W, Shuai Z, Jiang Y, Liu Y, Lipsky PE, Chen H; YISTAR study group. Efficacy and safety of tripterygium wilfordii Hook F plus TNF inhibitor for active rheumatoid arthritis: A multicentre, randomized, double-blind, triple-dummy controlled trial. Clin Immunol. 2023 Oct;255:109749. doi: 10.1016/j.clim.2023.109749. Epub 2023 Aug 30. PMID 37657525